CLINICAL TRIAL: NCT01144078
Title: Exercise Intensity, Glycemic Control and Abdominal Fat in People With Type 2 Diabetes: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Diabetes Institute (Other)
Responsible Party: Principal Investigator, Normand Boule, PhD, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADI-2010
Record Dates: First submitted 2010-06-07; First posted 2010-06-15 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Adiposity; Exercise training; Older adults
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity Interval Exercise (Experimental): This arms receives the High Intensity Interval Exercise intervention
  Interventions: Behavioral: High Intensity Interval Exercise
- Traditional Intensity Exercise (Experimental): This arms receives the Traditional Intensity Exercise intervention
  Interventions: Behavioral: Traditional Intensity Exercise

INTERVENTIONS:
Behavioral: Traditional Intensity Exercise — The exercise intensity will be set at a workload corresponding to 40% of the workload obtained at VO2peak during the baseline progressive maximal exercise tests. Based on the anticipated fitness of the participants this should to an intensity of about 3.5 METs, which is similar to walking at a moderate pace.
  Other Names: Low Intensity Exercise; Moderate Intensity Exercise
  Arms: Traditional Intensity Exercise
Behavioral: High Intensity Interval Exercise — The High Intensity Interval Exercise intervention will replicate all aspects of the Traditional Intensity Exercise with the exception of exercise intensity. The High Intensity Interval Exercise protocol will involve alternating between 1-minute intervals at 100% workload obtained at VO2peak followed by 3-minute recovery intervals at 20% of workload obtained at VO2peak (average = 40% ). As many complete intervals as possible will be completed during a training session (e.g., 7 intervals can be completed in a 30 min period (7 x 4 min = 28 min), with the remaining time spent at 40% peak workload to ensure a similar work output as the Traditional Intensity Exercise.
  Arms: High Intensity Interval Exercise

SUMMARY:
Body fat is an important risk factors for type 2 diabetes. However, not all body fat is the same. Research suggests that fat stored in the abdomen is most harmful. This is known as intra-abdominal fat. The objective of the proposed study is to understand the effect of exercise intensity on intra-abdominal fat and glucose control. Twenty participants with type 2 diabetes will be assigned to traditional or high intensity exercise. The exercise interventions will last a total of 14 weeks. Those in the traditional intensity group will exercise at an intensity comparable to walking. The high intensity group will alternate between 1 minute at high intensity and 3 minutes at low intensity. Both exercise groups will burn a similar amount of Calories and will exercise for the same amount of time. The exercise duration will start at 30 minutes per day. By the end of the study, it will be 60 minutes per day. All exercise sessions will be supervised. Body fat distribution will be estimated by a scanning machine called a DXA and anthropometric measures. Glycemic control will be measured from a blood sample. This study may not be of sufficient size to detect meaningful changes in these variables. However, it will provide information in regards to the preliminary efficacy, resource requirements and feasibility. Feasibility will include: recruitment, retention and adherence. Such information is essential for planning a more definitive trial. The identification of exercises that target greater reductions in abdominal fat will have important implications for the health of people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with type 2 diabetes.
* From 55-75 years of age (Women post-menopausal for at least 5 years).
* Sedentary: < 3 bouts of planed physical activity of >30 min per week.

Exclusion Criteria:

* Smoking (defined as more than one cigarette per day).
* Inability to speak and read English.
* Diseases known to affect body fat distribution (e.g., polycystic ovary syndrome, Cushing's syndrome, HIV-AIDS or lipodystrophies).
* Taking medications that may affect body fat distribution (e.g., Thiazolidinedione, Insulin, Growth Hormone).
* Limitations to regular exercise training (e.g., musculoskeletal limitations, heart disease, chronic obstructive pulmonary disease).
* Answering "yes" to any of the questions on the physical activity readiness questionnaire (PAR-Q).
* Having undergone major changes in physical activity, diet or medication in the previous 6 months (or be planning such changes in the next 4 months). Changes in physical activity will be considered as an increase or decrease of more than 1 hour per week. A change in body weight greater 3 kg will also lead to exclusion.
* Body weight > 300 lbs (maximum weight for Dual Energy X-Ray Absorptiometry (DXA) table).
* HbA1c > 0.09%
* blood pressure above 140/90 mmHg.
* LDL cholesterol above 3.5 mmol/L or TC:HDL-C above 5.0.
* Self-reported alcohol or substance abuse within the past twelve months, current consumption of more than 14 alcoholic drinks per week, and/or current acute treatment or rehabilitation program for these problems.
* Other medical or psychiatric factors that in the judgment of the principal investigators may interfere with study participation or the ability to follow the study protocol.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of these exercise interventions in people with type 2 diabetes | The feasibility of recruiting will be assessed over the 12-month recruitment phase. Adherence will be measured throughout the 14-week interventions. Retention will consider those who participate in the assessments before and after the intervention.
  * Recruitment
  * Adherence
  * Retention

SECONDARY OUTCOMES:
Intra-abdominal fat | During the week before and the week after the 14 week exercise interventions
  Intra-abdominal fat will be estimated by previously validated technique of combining DXA and anthropometric measurements (Bertin 2000)
Glycated hemoglobin (A1c) | During the week before and the week after the 14 week exercise interventions
Glucose | Before and after individual exercise sessions
  Throughout the intervention period, we will take regular capillary blood glucose and lactate measures with a OneTouch® Ultra (LifeScan; Milpitas, CA, USA) portable glucose analyzer and a Accusport® (Boehringer Mannheim, Castle Hill, Australia) portable lactate analyzer. Samples will be taken 5 minutes before and 5 minutes after the exercise bout.
Plasma lipids and lipoproteins | During the week before and the week after the 14 week exercise interventions
  * HDL cholesterol
  * LDL cholesterol
  * Total cholesterol
  * Triglycerides
Daily steps | During the week before the 14 week exercise interventions as well as during week 8 and week 14 of the interventions
  Daily steps will be measured with a Yamax SW-200Digiwalker Pedometer.
Dietary intake | During the week before the 14 week exercise interventions as well as during week 8 and week 14 of the interventions
  Dietary intake will be estimated by a standard 3-day food record (2 weekdays and 1 weekend).
Anthropometrics | During the week before and the week after the 14 week exercise interventions
  Anthropometrics will include: height, weight, waist circumference and hip circumference.
Blood pressure | During the week before and the week after the 14 week exercise interventions
Fitness | During the week before and the week after the 14 week exercise interventions
  A graded maximal cycle ergometer test will be conducted on a cycle ergometer. The test will begin at a pedal rate of 60-65 rpm and a resistance of 0 kp. Pedaling rate will remain constant but resistance will increase by 0.5 kp every 2 min until exhaustion. Respiratory gases will be analyzed throughout (TrueMax; ParvoMedics, Salt Lake City, UT, USA). Heart rate was continuously monitored with a polar heart rate monitor (Polar Electro, NY, USA).
Exercise Self-efficacy | During week 1, week 8 and week 14 of the exercise interventions
  A series of questions will be used to obtain preliminary information on the acceptability of the exercise protocols to the participants. The questions will include rating of perceived exertion (Borg Scale), as well as several indications of the participants confidence in being able to complete such exercise on a regular basis, including coping, task and scheduling self-efficacy. Other questions that related to fatigue will also be asked.

CONTACTS AND LOCATIONS:
Overall Officials: Normand G. Boulé, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Terada T, Friesen A, Chahal BS, Bell GJ, McCargar LJ, Boule NG. Exploring the variability in acute glycemic responses to exercise in type 2 diabetes. J Diabetes Res. 2013;2013:591574. doi: 10.1155/2013/591574. Epub 2013 Jul 29. PMID 23984433
- [Derived] Terada T, Friesen A, Chahal BS, Bell GJ, McCargar LJ, Boule NG. Feasibility and preliminary efficacy of high intensity interval training in type 2 diabetes. Diabetes Res Clin Pract. 2013 Feb;99(2):120-9. doi: 10.1016/j.diabres.2012.10.019. Epub 2012 Nov 24. PMID 23183390